CLINICAL TRIAL: NCT04246619
Title: Efficacy of Pregabalin and Duloxetine in Patients With Painful Diabetic Peripheral Neuropathy (PDPN): the Effect of Pain on Cognitive Function, Sleep and Quality of Life (BLOSSOM)
Brief Title: Efficacy of Pregabalin and Duloxetine in Patients With PDPN: the Effect of Pain on Cognitive Function, Sleep and Quality of Life
Acronym: BLOSSOM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The statistical analysis will still provide relevant results with the same statistical power as initially planned.COVID-19 pandemic prolonged the recruiting period and consequently affected the costs of the clinical trial.
Sponsor: KRKA (Industry)
Collaborators: 3ARH (Unknown); INTERBORA (Unknown); University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KCT 11/2017; 2017-004341-24 (EudraCT Number)
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Painful Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Pregabalin; Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Treatment is started at Visit 2 with Pregabalin Krka or Dulsevia - according to randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin Krka Arm (Experimental): ARM 1: pregabalin (Pregabalin Krka 25-150 mg/ day) FLEXIBLE-DOSE REGIMEN.
  Investigator can choose on V2:
  * Total Pregabalin Krka daily dose: 25 mg/day
  * Total Pregabalin Krka daily dose: 50 mg/day
  * Total Pregabalin Krka daily dose: 75 mg/day
  * Total Pregabalin Krka daily dose: 150 mg/day
  * Total Pregabalin Krka daily dose: 300 mg/day (from Phone call 1 further on)
  V3: daily dose should be achieved: MINIMUM dose 150 mg/day Investigator can choose: total Pregabalin Krka daily dose 150 mg/day or 300 mg/day or 600 mg/day Investigator can choose: total Pregabalin Krka daily dose 150 mg/day or 300 mg/day or 600 mg/day
  V4: Investigator can choose: total Pregabalin Krka daily dose 150 mg/day or 300 mg/day or 600 mg/day
  Interventions: Drug: Pregabalin
- Dulsevia® Arm (Experimental): • ARM 2: duloxetine (Dulsevia® 30-60 mg/ day) FLEXIBLE-DOSE REGIMEN:
  Investigator can choose on V2:
  * Total Dulsevia® daily dose: 30 mg/day
  * Total Dulsevia® daily dose: 60 mg/day
  V3: daily dose should be achieved: MINIMUM dose 60 mg/day Investigator can choose total Dulsevia® daily dose 60 mg/day or 90 mg/day or 120 mg/day.
  V4: Investigator can choose total Dulsevia® daily dose 60 mg/day or 90 mg/day or 120 mg/day.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Pregabalin — Pregabalin Krka (pregabalin) hard capsules of different strenghts: 25 mg, 75 mg, 150 mg, 300 mg.
  Duration: 12 weeks
  Arms: Pregabalin Krka Arm
Drug: Duloxetine — Dulsevia® (duloxetine) hard gastro-resistant capsules of different strenghts: 30 mg and 60 mg.
  Duration: 12 weeks
  Arms: Dulsevia® Arm

SUMMARY:
The objective and the purpose of the trial is to: assess the efficacy of Pregabalin Krka and Dulsevia® in patients with PDPN, investigate the effect of Pregabalin Krka and Dulsevia® on pain and on quality of life (QOL), depression symptoms, cognitive functions, sleep quality and daytime sleepiness and assess the safety of Pregabalin Krka and Dulsevia® in patients with PDPN.

During the 3 months (12 weeks) 5 visits and 2 phone calls are planned.

After the ICF signature and before therapy is allocated, a screening procedure is carried out to verify eligibility: laboratory analyses (concentrations of TSH, vitamin B12, folic acid, glucose, HbA1c, pregnancy test for women of childbearing potential), assessment of PDPN (with questionnaire DN4), assessment of cognition (with questionnaire MoCA), habits, medical history (medical/surgical history and concomitant diseases, previous and/or existing therapy of pain in PDPN, concomitant medications) with measurements and evaluation of pain according to VAS.

On Visit 2 investigator checks the results of laboratory tests, of pregnancy test, measures vital signs, evaluates pain in PDPN according to VAS, checks previous analgesic therapy and concomitant medications.

If patient meets all inclusion and exclusion criteria, he/she is eligible and will be randomly assigned (automatically through electronic version of case report form (eCRF) into two therapy groups (treatment arms) - tretament with Pregabalin Krka OR treatment with Dulsevia®.

Investigator performs assessments of: QoL, sleep quality and daytime sleepiness, depression and adverse events.

At Visit 3, compliance monitoring is done, pain intensity in PDPN by VAS is evaluated, concomitant therapy is checked, vital signs are measured, doses of IMP are adjusted and adverse events assessment are carried out.

At Visit 4, pregnancy test for women of childbearing potential and compliance monitoring are carried out; concomitant medications are checked, vital signs are measured, pain intensity in PDPN by VAS is evaluated, IMP are adjusted and assessment of adverse events is carried out.

At Visit 5 investigator performs again assessments of: QoL, sleep quality and daytime sleepiness, depression, cognition and PDPN. Evaluation of the pain intensity in PDPN by VAS and assessment of the adverse events should be performed. Pregnancy test for women of childbearing potential is carried out.

DETAILED DESCRIPTION:
During the 3 months (12 weeks) 5 visits and 2 phone calls are planned.

Procedures and administration:

On arrival at the trial site at Visit 1 the patient receives the complete information on the trial procedures. The patient confirms his decision to participate by signing the informed consent form (ICF). After the ICF signature and before therapy is allocated, a screening procedure is carried out to verify eligibility: laboratory analyses (concentrations of TSH, vitamin B12, folic acid, glucose, HbA1c, pregnancy test for women of childbearing potential), assessment of PDPN (with questionnaire DN4), assessment of cognition (with questionnaire MoCA), habits, medical history (medical/surgical history and concomitant diseases, previous and/or existing therapy of pain in PDPN, concomitant medications) with measurements and evaluation of pain according to VAS.

Patient is instructed not to take any PDPN medication and/or analgesics, if existing on a day of Visit 2.

Information obtained at Visit 1 is input in the eCRF.

Visit 2 (initial baseline visit): 0-7 days after Visit 1

Investigator checks the results of laboratory tests, of pregnancy test, measures vital signs (heart rate, blood pressure), evaluates pain in PDPN according to VAS (separate assessments of current pain intensity, average pain intensity in last 24-h, worst pain intensity in last 24-h, average pain intensity in last 4 weeks and worst pain intensity in last 4 weeks), checks previous analgesic therapy and concomitant medications.

If patient meets all inclusion and exclusion criteria, he/she is eligible and will be randomly assigned (automatically through electronic version of case report form (eCRF) into two therapy groups (treatment arms).

Investigator performs assessments of: QoL (with questionnaire SF-36), sleep quality and daytime sleepiness (with questionnaires ISI and ESS), depression (with questionnaire MDI) and adverse events.

Administration:

Eligible screened patients are randomly assigned into two therapy groups (treatment arms):

ARM 1: treatment with pregabalin (Pregabalin Krka) or ARM 2: treatment with duloxetine (Dulsevia®).

Each patient receives a Patient diary number 1, including the doses of Pregabalin Krka or Dulsevia® (depending on randomization) from Visit 2 (day 1) till Phone call 1, scales for assessing the pain and with the date of Phone call 1.

Treatment during PERIOD 1 (FLEXIBLE-DOSE REGIMEN during the first 14 days (±3 days) in order to allow the investigator to give each patient an optimal dose of IMP.

* ARM 1: pregabalin (Pregabalin Krka 25-150 mg/ day) FLEXIBLE-DOSE REGIMEN. Investigator can choose total Pregabalin Krka daily dose: 25 mg/day, 50 mg/day, 75 mg/day, 150 mg/day or 300 mg/day (from Phone call 1 further on)
* ARM 2: duloxetine (Dulsevia® 30-60 mg/ day) FLEXIBLE-DOSE REGIMEN:

Investigator can choose total Dulsevia® daily dose: 30 mg/day or 60 mg/day

At the Visit 2, RM is given to each patient to cover the treatment till the next Visit 3.

Phone call 1: week 1 (± 3 days) At week 1 (7 ± 3 days after Visit 2) investigator calls the patient by phone and ask him or her about possible adverse events and to evaluate the pain intensity in PDPN by VAS which is a part of Patient diary 1.

Investigator can adjust the dose of IMP during phone call:

* If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) is NOT achieved, the investigator can increase the dose;
* if bothersome adverse event occurs the investigator can decrease the dose (if possible).

The investigator also ask the patient if he or she is taking the IMP appropriately (according to investigator's instructions).

NOTE: On the next visit (Visit 3; 14 ± 3 days after Visit 2) following daily doses should be achieved by each patient:

* ARM 1: Total Pregabalin Krka daily dose: MINIMUM dose 150 mg/day
* ARM 2: Total Dulsevia daily dose: MINIMUM dose 60 mg/day

Visit 3: week 2 (14 ± 3 days after Visit 2) At Visit 3, compliance monitoring is done, pain intensity in PDPN by VAS is evaluated, concomitant therapy is checked, vital signs are measured, doses of IMP are adjusted and adverse events assessment are carried out.

Investigator collects the Patient Diary 1. Data in Patient Diary 1 are checked.Treatment during PERIOD 2 (it lasts 6 weeks)

Treatment options:

ARM 1: pregabalin (Pregabalin Krka) Investigator can choose: total Pregabalin Krka daily dose: 150 mg/day or 300 mg/day or 600 mg/day

NOTE:

If in the opinion of the investigator the minimum IMP dose of 150 mg of Pregabalin Krka/ 60 mg of Dulsevia® can not be reached after Visit 3, the patient must be excluded from the trial.

ARM 2: duloxetine (Dulsevia®)

Investigator can choose:

* total Dulsevia® daily dose*: 60 mg/day or 90 mg/day* or total Dulsevia® daily dose**: 120 mg/day

  * once daily dosing by using available dosages. **the daily dose will be achieved with two devided doses of Dulsevia® by using available dosages.

ARM 1: pregabalin (Pregabalin Krka)

* If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with baseline is achieved during period 1, further treatment with Pregabalin Krka 150 mg/day or 300 mg/day in the period 2 is required.
* If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with baseline is NOT achieved, further treatment with a dose of:

  * 150 mg/day (if patient was till now treated with equal dose) or 300 mg/day (if patient was till now treated with equal dose to 150 mg or 300 mg) or 600 mg/day (if patient was till now treated with equal dose to 300 mg) is required.

ARM 2: duloxetine (Dulsevia®)

* If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with baseline is achieved further treatment with Dulsevia® 60 mg/day in the period 2 is required.
* If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with baseline is NOT achieved, further treatment with the dose of:

  * Dulsevia® 60 mg/day (if patient was till now treated with equal dose) or Dulsevia® 90 mg/day (if patient was till now treated with lower dose) or Dulsevia® 120 mg/day (if patient was till now treted with lower dose) is required.

At the Visit 3, RM is given to each patient to cover the treatment till the next Visit 4. Patient is requested to bring packages with all blisters (empty blisters and blister with unused IMPs and RM) on the Visit 4.

Each patient receives a Patient diary number 2, including the doses of Pregabalin Krka or Dulsevia® (depending on randomization) from Visit 3 till Phone call 2, scales for assessing the pain and with the date of Phone call 2 (28 ± 3 days after Visit 3).

Patient is requested to bring the Patient diary on the next visit.

Information obtained at Visit 3 is input in the eCRF.

Phone call 2: 4 weeks(28 ± 3 days) after visit 3 At week 6 (28 ± 3 days after Visit 3) the investigator again calls the patient by phone and asks him or her about possible bothersome adverse events and to evaluate the pain intensity in PDPN by VAS (separate assessments of current pain intensity, average pain intensity in last 24-h and worst pain intensity in last 24-h) which is a part of Patient diary 2.

The investigator can adjust the dose of Pregabalin Krka or Dulsevia®, if necessary. If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) is NOT achieved the investigator can increase the dose and if bothersome adverse event occurs the investigator can decrease the dose to the previous dose.

The investigator also checks if the patient takes the medicines appropriately (according to investigator's instructions).

Visit 4: week 8 (42 ± 3 days after Visit 3) At Visit 4, pregnancy test for women of childbearing potential and compliance monitoring are carried out; concomitant medications are checked, vital signs are measured, pain intensity in PDPN by VAS is evaluated (separate assessments of current pain intensity, average pain intensity in last 24-h and worst pain intensity in last 24-h, average pain intensity in last 4 weeks and worst pain intensity in last 4 weeks), IMP are adjusted and assessment of adverse events is carried out. Investigator collects the Patient Diary 2. Data in Patient Diary 2 are checked.

Treatment options during PERIOD 3 (it lasts 4 weeks) ARM 1: pregabalin (Pregabalin Krka)

Investigator can choose:

Total Pregabalin Krka daily dose: 75 mg/day *,150 mg/day, 300 mg/day or 600 mg/day

*only in case of bothersome adverse events

ARM 2: duloxetine (Dulsevia®) Investigator can choose:Total Dulsevia® daily dose: 30 mg/day*, 60 mg/day, 90 mg/day or 120 mg/day *only in case of bothersome adverse events

Arm 1: pregabalin (Pregabalin Krka)

• If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with Visit 3 is achieved, further treatment with previous dose in the period 3 is required.

• If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with Visit 3 is NOT achieved on daily dose 150 mg, further treatment with a dose of: 150 mg/day (if patient was till now treated with equal dose) or 300 mg/day (if patient was till now treated with lower or equal dose) or 600 mg/day (if patient was till now treted with lower or equal dose) is required.

Arm 2: duloxetine (Dulsevia®)

* If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with Visit 3 is achieved further treatment with previous dose in the period 3 is required.
* If average pain intensity in PDPN in last 24-h equal or below 30 mm (measured by VAS) or reduction of pain equal or more than 30 % compared with Visit 3 is NOT achieved, further treatment with a dose of:

Dulsevia® 60 mg/day (if patient was till now treated with equal dose) or Dulsevia® 90 mg/day (if patient was till now treated with lower or equal dose) or Dulsevia® 120 mg/day (if patient was till now treated with lower or equal dose).

At the Visit 4, RM is given to each patient to cover the treatment till the next Visit 5.

Visit 5: week 12 (28 ± 3 days after Visit 4) At Visit 5 investigator performs again assessments of: QoL, sleep quality and daytime sleepiness, depression, cognition and PDPN.

Evaluation of the pain intensity in PDPN by VAS and assessment of the adverse events should be performed.

Pregnancy test for women of childbearing potential is carried out.

Compliance monitoring, measurement of vital signs and concomitant medications are also carryed out by investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients aged 18-85 years.
2. Patients with a history of type 2 diabetes mellitus according to The American Diabetes Association (ADA).
3. Patients with a diagnosis of painful diabetic peripheral neuropathy (PDPN) caused by type 2 diabetes mellitus based on DN4 ≥4.
4. Patients whose average pain intensity in PDPN in last 24 hours (measured by VAS), evaluated on baseline visit, is equal or more than 40 mm (0 mm ='no pain' and 100 mm ='worst possible pain').
5. Ability to adhere to trial protocol.
6. Written informed consent.

The methods for inclusion criteria assessment include medical history, interview, completing the DN4 questionnaire, physical examination, assesment of pain on VAS and laboratory analyses.

Exclusion Criteria:

1. Patients who took PDPN medication and/or analgesics on a day of baseline visit.
2. Patients with a known hypersensitivity to duloxetine, pregabalin, paracetamol or tramadol or any of the inactive ingredients or have any contraindication for the use of duloxetine, pregabalin, paracetamol or tramadol.
3. Patients with a history of inadequate pain response (pain reduced was equal or less than 30%) to:

   3.1. pregabalin at maximum allowed treatment daily dose 600 mg, 3.2. duloxetine at maximum allowed treatment daily dose 120 mg, 3.3. venlafaxine at maximum allowed treatment daily dose 375 mg, 3.4. gabapentin on daily treatment dose more than 1800 mg 3.5. amitriptilin at maximum allowed treatment daily dose 150 mg.
4. Patients, who are currently treated with a daily dose that exceeds:

   4.1. 150 mg of pregabalin, 4.2. 60 mg of duloxetine, 4.3. 150 mg of venlafaxine, 4.4. 600 mg of gabapentin.
5. Patients with an uncontrolled type 2 diabetes mellitus.
6. The average scores of less than 20 on MoCA.
7. Have any other type of neuropatic pain, contrasted to PDPN.
8. Evidence of another cause of distal polyneuropathy other than diabetic.
9. Have a serious (evaluated by physician) unstable cardiovascular (e.g. uncontrolled hypertension), hepatic, renal, respiratory, ophthalmologic, gastrointestinal, or hematologic illness, symptomatic peripheral vascular disease, malignant disease or other medical condition that could lead to hospitalisation during the course of the trial.
10. Have a diagnosis or history of uncontrolled glaucoma.
11. Known or suspected alcohol or drug abuse or addiction (excluding nicotine and caffeine).
12. Patients with a history of depression (less than one year after completing the last medical treatment), mania, bipolar disorder, psychosis or schizophrenia.
13. Pregnancy, lactation and women of child-bearing potential without highly effective* or at least acceptable** contraception (according to the Recommendations related to contraception and pregnancy testing in clinical trials).
14. Patients with a history of epilepsy, stroke or neurodegenerative disease.
15. Patients taking Monoamine oxidase (MAO) inhibitors or are within one year of their withdrawal.
16. Acute liver injury (such as hepatitis) or severe cirrhosis (Child-Pugh Class C).
17. Patients with suspected Restless leg syndrome (RLS).
18. Abnormal thyroid-stimulating hormone (TSH) concentrations (according to the references value of the local laboratory).
19. Vitamin B12 and folic acid deficiency (according to the reference values of the local laboratory).
20. Surgical procedures planned to occur during trial (patients may be rescreened following completion of and recovery from the surgical procedure).
21. Concomitant treatment that might influence the final therapeutic effect of the tested active substances including non-medical treatments.
22. Patients who under the opinion of the investigator will not be compliant to the treatment or not be able to finish the trial for any other reason.

    * Highly effective contraception is:

      * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation(oral, intravaginal, transdermal)
      * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
      * intrauterine device (IUD)
      * intrauterine hormone-releasing system (IUS)
      * bilateral tubal occlusion
      * vasectomised partner
      * sexual abstinence

        **Acceptable contraception is:
      * progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
      * male or female condom with or without spermicide
      * cap, diaphragm or sponge with spermicide

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Clinically meaningful improvement of pain in PDPN after a 12 week treatment with pregabalin | 12 weeks
  Clinically meaningful improvement of pain in PDPN after a 12 week treatment according to VAS
Clinically meaningful improvement of pain in PDPN after a 12 week treatment with duloxetine | 12 weeks
  Clinically meaningful improvement of pain in PDPN after a 12 week treatment according to VAS

SECONDARY OUTCOMES:
The proportion of patients with reduction of pain in PDPN for equal or more than 30 % AND/OR with pain intensity in PDPN not exceeding 30 mm | week 1, week 2, week 6, week 8
  The proportion of patients with reduction of pain in PDPN (measured by VAS) for equal or more than 30 % AND/OR with pain intensity in PDPN not exceeding 30 mm (measured by VAS) taking into consideration:
  i. current pain intensity (measured at doctor's office)
  ii. average pain intensity in last 24-h
  iii. worst pain intensity in last 24-h
The proportion of patients with reduction of pain in PDPN for equal or more than 30 % AND/OR with pain intensity in PDPN not exceeding 30 mm | week 8, week 12
  The proportion of patients with reduction of pain in PDPN for equal or more than 30 % (measured by VAS) AND/OR with pain intensity in PDPN not exceeding 30 mm (measured by VAS) taking into consideration:
  i. average pain intensity in last 4 weeks
  ii. worst pain intensity in last 4 weeks
Pain intensity difference in PDPN | week 1, week 2, week 6, week 8, week 12
  Pain intensity difference in PDPN (measured by VAS) between each control visit/ phone call and the baseline value at Visit 2:
  i. current pain intensity (measured at doctor's office)
  ii. average pain intensity in last 24-h
  iii. worst pain intensity in last 24-h
Pain intensity difference in PDPN | week 8, week 12
  Pain intensity difference in PDPN (measured by VAS) between Visits 4 and 5 and the baseline value at Visit 2:
  i. average pain intensity in last 4 weeks
  ii. worst pain intensity in last 4 week
The proportion of patients with reduction of pain in PDPN for equal or more than 50 % | Baseline vs.: week 1, week 2, week 6, week 8, week 12
  The proportion of patients with reduction of pain in PDPN (measured by VAS) for equal or more than 50 % taking into consideration:
  i. current pain intensity (measured at doctor's office)
  ii. average pain intensity in last 24-h
  iii. worst pain intensity in last 24-h
The proportion of patients with reduction of pain in PDPN for equal or more than 50 % | week 8, week 12
  The proportion of patients with reduction of pain in PDPN (measured by VAS) for equal or more than 50 % taking into consideration:
  i. average pain intensity in last 4 weeks
  ii. worst pain intensity in last 4 weeks
The proportion of patients with eliminated pain in PDPN | week 6, week 8, week 12
  The proportion of patients with eliminated pain in PDPN, which includes intensity of pain in PDPN not exceeding 10 mm (measured by VAS) taking into consideration:
  i. current pain intensity (measured at doctor's office)
  ii. average pain intensity in last 24-h
  iii. worst pain intensity in last 24-h
The proportion of patients with eliminated pain in PDPN | week 8, week 12
  The proportion of patients with eliminated pain in PDPN, which includes intensity of pain in PDPN not exceeding 10 mm (measured by VAS) taking into consideration:
  i. average pain intensity in last 4 weeks
  ii. worst pain intensity in last 4 weeks
Dose-related efficacy | week 2, week 8, week 12
  Changes of efficacy according to changing of doses
DN4 score difference | baseline, week 12
  Mean changes of scores
Quality of life (QoL) difference with 36-Item Short Form Survey Instrument (SF-36) | baseline, week 12
  Mean changes of scores
The Montreal Cognitive Assessment (MoCA) score difference for cognitive improvement | week 1, week 12
  Mean changes of scores
Insomnia severity index (ISI) difference for sleep | baseline, week 12
  Mean changes of scores
Epworth Sleepiness Scale (ESS) score for daytime sleepiness improvement | baseline, week 12
  Mean changes of scores
Major depression inventory (MDI) score difference for improvement of major depression | baseline, week 12
  Mean changes of scores
Proportion of compliant patients | week 2, week 8, week 12
  Proportion of compliant patients, i.e. those having a compliance of more than 80 % at the regular therapy end visit

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rakuša, Study Chair — University Medical Centre Maribor
Locations (13):
- Croatia (4):
  - Opća bolnica Karlovac, Karlovac
  - Clinical Medical Center Osijek, Osijek
  - KB Merkur, Sveučilišna klinika Vuk Vrhovac, Zagreb
  - Klinička bolnica Sveti Duh, Zagreb
- North Macedonia (2):
  - JZU Univerzitetska klinika za endokrinologija, dijabetes I metabolicki bolesti - Skopje, Skopje
  - JZU Univerzitetska klinika za nevrologija, Skopje
- Poland (2):
  - Gabinet Neurologiczny, prof. Adam Stępień, Warsaw
  - Poradnia neurologiczna, Centrum terapii dzieci i Dorosłych FIMEDICA Sp. z o.o., Warsaw
- Serbia (3):
  - Klinički centar Srbije, Belgrade
  - Klinički centar Niš, Niš
  - Klinički centar Vojvodine, Novi Sad
- Slovenia (2):
  - Zdravstveni dom Koper, Koper
  - Clemenz Marjetka - Nevrološka Ordinacija, Ljubljana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Menachem E. Pregabalin pharmacology and its relevance to clinical practice. Epilepsia. 2004;45 Suppl 6:13-8. doi: 10.1111/j.0013-9580.2004.455003.x. PMID 15315511
- [Background] Tassone DM, Boyce E, Guyer J, Nuzum D. Pregabalin: a novel gamma-aminobutyric acid analogue in the treatment of neuropathic pain, partial-onset seizures, and anxiety disorders. Clin Ther. 2007 Jan;29(1):26-48. doi: 10.1016/j.clinthera.2007.01.013. PMID 17379045
- [Background] Schulze-Bonhage A. Pharmacokinetic and pharmacodynamic profile of pregabalin and its role in the treatment of epilepsy. Expert Opin Drug Metab Toxicol. 2013 Jan;9(1):105-15. doi: 10.1517/17425255.2013.749239. Epub 2012 Dec 4. PMID 23205518
- [Background] Bockbrader HN, Wesche D, Miller R, Chapel S, Janiczek N, Burger P. A comparison of the pharmacokinetics and pharmacodynamics of pregabalin and gabapentin. Clin Pharmacokinet. 2010 Oct;49(10):661-9. doi: 10.2165/11536200-000000000-00000. PMID 20818832
- [Background] Goldstein DJ. Duloxetine in the treatment of major depressive disorder. Neuropsychiatr Dis Treat. 2007 Apr;3(2):193-209. doi: 10.2147/nedt.2007.3.2.193. PMID 19300553
- [Background] Perahia DG, Pritchett YL, Desaiah D, Raskin J. Efficacy of duloxetine in painful symptoms: an analgesic or antidepressant effect? Int Clin Psychopharmacol. 2006 Nov;21(6):311-7. doi: 10.1097/01.yic.0000224782.83287.3c. PMID 17012978
- [Background] Lesser H, Sharma U, LaMoreaux L, Poole RM. Pregabalin relieves symptoms of painful diabetic neuropathy: a randomized controlled trial. Neurology. 2004 Dec 14;63(11):2104-10. doi: 10.1212/01.wnl.0000145767.36287.a1. PMID 15596757
- [Background] Rosenstock J, Tuchman M, LaMoreaux L, Sharma U. Pregabalin for the treatment of painful diabetic peripheral neuropathy: a double-blind, placebo-controlled trial. Pain. 2004 Aug;110(3):628-638. doi: 10.1016/j.pain.2004.05.001. PMID 15288403
- [Background] Richter RW, Portenoy R, Sharma U, Lamoreaux L, Bockbrader H, Knapp LE. Relief of painful diabetic peripheral neuropathy with pregabalin: a randomized, placebo-controlled trial. J Pain. 2005 Apr;6(4):253-60. doi: 10.1016/j.jpain.2004.12.007. PMID 15820913
- [Background] Tolle T, Freynhagen R, Versavel M, Trostmann U, Young JP Jr. Pregabalin for relief of neuropathic pain associated with diabetic neuropathy: a randomized, double-blind study. Eur J Pain. 2008 Feb;12(2):203-13. doi: 10.1016/j.ejpain.2007.05.003. Epub 2007 Jul 16. PMID 17631400
- [Background] Razazian N, Baziyar M, Moradian N, Afshari D, Bostani A, Mahmoodi M. Evaluation of the efficacy and safety of pregabalin, venlafaxine, and carbamazepine in patients with painful diabetic peripheral neuropathy. A randomized, double-blind trial. Neurosciences (Riyadh). 2014 Jul;19(3):192-8. PMID 24983280
- [Background] Freynhagen R, Strojek K, Griesing T, Whalen E, Balkenohl M. Efficacy of pregabalin in neuropathic pain evaluated in a 12-week, randomised, double-blind, multicentre, placebo-controlled trial of flexible- and fixed-dose regimens. Pain. 2005 Jun;115(3):254-263. doi: 10.1016/j.pain.2005.02.032. Epub 2005 Apr 18. PMID 15911152
- [Background] Lindsay TJ, Rodgers BC, Savath V, Hettinger K. Treating diabetic peripheral neuropathic pain. Am Fam Physician. 2010 Jul 15;82(2):151-8. PMID 20642268
- [Background] Goldstein DJ, Lu Y, Detke MJ, Lee TC, Iyengar S. Duloxetine vs. placebo in patients with painful diabetic neuropathy. Pain. 2005 Jul;116(1-2):109-18. doi: 10.1016/j.pain.2005.03.029. PMID 15927394
- [Background] Raskin J, Pritchett YL, Wang F, D'Souza DN, Waninger AL, Iyengar S, Wernicke JF. A double-blind, randomized multicenter trial comparing duloxetine with placebo in the management of diabetic peripheral neuropathic pain. Pain Med. 2005 Sep-Oct;6(5):346-56. doi: 10.1111/j.1526-4637.2005.00061.x. PMID 16266355
- [Background] Wernicke JF, Pritchett YL, D'Souza DN, Waninger A, Tran P, Iyengar S, Raskin J. A randomized controlled trial of duloxetine in diabetic peripheral neuropathic pain. Neurology. 2006 Oct 24;67(8):1411-20. doi: 10.1212/01.wnl.0000240225.04000.1a. PMID 17060567
- [Background] Raskin J, Wang F, Pritchett YL, Goldstein DJ. Duloxetine for patients with diabetic peripheral neuropathic pain: a 6-month open-label safety study. Pain Med. 2006 Sep-Oct;7(5):373-85. doi: 10.1111/j.1526-4637.2006.00207.x. PMID 17014595
- [Background] Wernicke JF, Raskin J, Rosen A, Pritchett YL, D'Souza DN, Iyengar S, Knopp K, Le TK. Duloxetine in the long-term management of diabetic peripheral neuropathic pain: An open-label, 52-week extension of a randomized controlled clinical trial. Curr Ther Res Clin Exp. 2006 Sep;67(5):283-304. doi: 10.1016/j.curtheres.2006.10.001. PMID 24678103
- [Background] Smith T, Nicholson RA. Review of duloxetine in the management of diabetic peripheral neuropathic pain. Vasc Health Risk Manag. 2007;3(6):833-44. PMID 18200804
- [Background] Wernicke JF, Prakash A, Kajdasz DK, Houston J. Safety and tolerability of duloxetine treatment of diabetic peripheral neuropathic pain between patients with and without cardiovascular conditions. J Diabetes Complications. 2009 Sep-Oct;23(5):349-59. doi: 10.1016/j.jdiacomp.2008.07.004. Epub 2008 Sep 2. PMID 18768332
- [Background] Attal N, Cruccu G, Baron R, Haanpaa M, Hansson P, Jensen TS, Nurmikko T. EFNS guidelines on the pharmacological treatment of neuropathic pain: 2010 revision. Eur J Neurol. 2010 Sep;17(9):1113-e88. doi: 10.1111/j.1468-1331.2010.02999.x. Epub 2010 Apr 9. PMID 20402746
- [Background] Shneker BF, McAuley JW. Pregabalin: a new neuromodulator with broad therapeutic indications. Ann Pharmacother. 2005 Dec;39(12):2029-37. doi: 10.1345/aph.1G078. Epub 2005 Nov 15. PMID 16288079
- [Background] Lunn MP, Hughes RA, Wiffen PJ. Duloxetine for treating painful neuropathy, chronic pain or fibromyalgia. Cochrane Database Syst Rev. 2014 Jan 3;2014(1):CD007115. doi: 10.1002/14651858.CD007115.pub3. PMID 24385423
- [Background] Del Casale A, Girardi P, Brugnoli R, Sani G, Di Pietro S, Brugnoli C, Caccia F, Angeletti G, Serata D, Rapinesi C, Tatarelli R, Kotzalidis GD. Duloxetine in the treatment of elderly people with major depressive disorder. Riv Psichiatr. 2012 Nov-Dec;47(6):479-88. doi: 10.1708/1178.13054. PMID 23160108
- [Derived] Rakusa M, Marolt I, Stevic Z, Rebrina SV, Milenkovic T, Stepien A. Efficacy of Pregabalin and Duloxetine in Patients with Painful Diabetic Peripheral Neuropathy (PDPN): A Multi-Centre Phase IV Clinical Trial-BLOSSOM. Pharmaceuticals (Basel). 2023 Jul 18;16(7):1017. doi: 10.3390/ph16071017. PMID 37513930